CLINICAL TRIAL: NCT00932724
Title: Phase II Double-blind Placebo-controlled Trial of CY503 in Patients With Chemotherapy-refractory Metastatic Colorectal Cancer
Brief Title: CY-503 for the Treatment of Chemotherapy-refractory Metastatic Colorectal Cancer
Acronym: CY503C2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor declared the early termination of the study due to poor recruitment of patients.
Sponsor: Cytavis Biopharma GmbH (Industry)
Collaborators: ClinAssess GmbH (Industry); Medical University Innsbruck (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Prof. Hans Lentzen, PhD, Cytavis Biopharma GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CY503C2; EudraCT no. 2008-005536-32
Record Dates: First submitted 2009-06-25; First posted 2009-07-03 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2011-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic; Colorectal; Cancer; refractory; Phase II; randomised; double-blind; controlled; multicenter; CY-503; Cytavis
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CY-503 (Experimental)
  Interventions: Drug: CY-503
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CY-503 — Ampoules with 1 ml 350 ng CY-503 solution for s.c. injection twice weekly. One cycle is defined as 4 consecutive weeks
  Arms: CY-503
Drug: Placebo — Ampoules with 1 ml placebo solution for s.c. injection twice weekly. One cycle is defined as 4 consecutive weeks
  Arms: Placebo

SUMMARY:
This trial is designed as a phase II evaluation of the effect of CY-503 or placebo on progression free survival (PFS) defined as the time from start of treatment until the objective observation of progressive disease (PD) or death from any course in patients with chemotherapy-refractory metastatic colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer has a worldwide annual incidence of approximately 1 million new cases diagnosed yearly and it is the second leading cause of cancer-related death in Western nations. There are a couple of approved standard therapies for the treatment of MCRC with cytotoxic agents irinotecan, oxaliplatin, and the fluoropyrimidines , as well as bevacizumab, the antibody against vascular endothelial growth factor A, and cetuximab, the antibody against the epidermal growth factor receptor. But there are only a few studies achieving a median survival time of more than 20 months in MCRC patients with standard regimens. After a 1st line therapy a high proportion (50% to 80%) of patients receives a 2nd line therapy with drugs not used in 1st line therapy and a part of them gets a 3rd line treatment. Results from a 2nd line therapy are best response rates ranging from 4 % - 23 %, a median PFS rate of 5.1 months, a median TTP of 4.1 - 4.6 months and median overall survival 6.9 - 12 months. However, for patients who experience disease progression after standard therapy (definition see inclusion criteria) there is no further standard therapeutic option. These patients developed a resistance to these therapies and finally die of their disease. They generally get best supportive care (BSC). Thus, there is a need for new active treatment options in this setting.

In this phase II double-blind placebo-controlled trial the efficacy and safety of CY-503, 350 ng s.c. injected in patients with chemotherapy refractory MCRC are tested. Approved treatments given to MCRC patients are usually discontinued after a treatment over some weeks at the first detection of objective PD. It will be tested if CY-503 is able to achieve progression-free-survival (PFS) in comparison to placebo. Patients will initially be included to receive either CY-503 or placebo until documentation of objective PD.

Standard therapy must be finished and has shown objective PD. Also patients with contraindications to standard therapy can be included.

CY-503 shows the potential to improve treatment of MCRC. This study aims at evaluating the activity and therapeutic effects of the substance. Anticipated capabilities are substitution of cytostatic drugs or improvement of their efficacy and tolerability . Furthermore, the expected improvement of PFS rates after failure of standard chemotherapies has to be investigated.

In a phase I trial CY-503 showed SD in patients who had exhausted standard therapy options for metastatic disease with subsequent disease progression with a median TTP of 17.4 weeks.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Patients are eligible with diagnosis of measurable metastatic colorectal carcinoma and radiologic documentation of disease progression during or with 3 months after termination of standard chemotherapy (fluoropyrimidine-based therapy with oxaliplatin and irinotecan). Patients who had to interrupt the 1st or 1nd line therapy due to intolerance or who were refractory or intolerant to the standard treatment regimens are eligible, too. Bevacizumab can, but does not need to be administered at discretion of treating physician. Patients with K-RAS wild-type can be treated with cetuximab or panitumumab before they enter the study.
* No chemotherapy within 4 weeks before treatment start
* No residual significant toxicity (greater than NCI grade 1), in case of peripheral neuropathy: no symptoms of peripheral neuropathy of NCI CTC grade 4 within 4 weeks before treatment start.
* No previous treatment with experimental therapies after standard therapies is allowed.
* Patients must use effective contraception if of reproductive potential. Females must not be pregnant or lactating
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 - 2
* WBC ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, platelet count ≥100,000/mm3
* Bilirubin ≤ 2.0 mg/dL (40 μmol/L) (unless due to Gilbert's syndrome in which case the bilirubin should be ≤3.5 mg/dL (59.86 μmol/L)), aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 5 × upper limit of normal (ULN); hepatic alkaline phosphatase ≤ 3.0 × ULN (in case of liver metastases higher levels do not hinder inclusion of patients)
* Serum creatinine ≤ 2.0 mg/dL (180 μmol/L)or creatinine clearance >= 50 ml/min. , proteinuria < 2.0 g/24 hr urine collection in patients with a positive urine dipstick for protein
* Written informed consent according to ICH-GCP and national laws and regulations prior to receipt of any trial medication or beginning trial procedures

Exclusion Criteria:

* Evidence of any other malignant disease (with the exception of tumors operatively cured at least 5 years prior to the trial)
* Known brain metastases
* Uncontrolled pleural effusions
* Interstitial pneumonitis or pulmonary fibrosis
* Severe/ unstable systemic disease or infection and circumstances not permitting trial participation (e.g., alcoholism or substance abuse)
* Unstable cardiac disease in the last 6 months
* Use of conventional mistletoe preparations, any immunostimulating substances and/or monoclonal antibodies within four weeks prior to and during the trial - ongoing therapy with steroids is permitted if the dose is not higher than 20 mg of prednisone-equivalent at the time of inclusion and during this clinical trial
* Any evidence or history (elicited by the investigator) of symptomatic cerebrovascular events (i.e., stroke or transient ischemic attack) within 6 months prior to randomization
* Any history or evidence of pulmonary embolism or thrombophlebitis (including deep vein thrombosis) requiring anticoagulant therapy (e.g., marcumar or heparin)
* History of hypersensitivity to mistletoe
* History of primary immunodeficiency
* Known human immunodeficiency virus (HIV) or known active viral hepatic infections
* Prior treatment with CY-503
* A general medical or psychological condition or behaviour, including substance dependence or abuse that, in the opinion of the investigator, might not permit the patient to complete the trial or sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Tumor assessment by using CT scans and/or MRIs | every 8 weeks (each 2 cycles)

SECONDARY OUTCOMES:
Assessment of Adverse Events | every 4 weeks (every cycle)
Assessment of quality of life using a standardized questionaire | every 4 weeks (every cycle)
Assessment of survival by "physical exam" | every 4 weeks (every cycle) / every 3 months during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Zwierzina, MD, Principal Investigator — University Hospital Innsbruck, Austria; Lothar Bergmann, MD, Principal Investigator — University Hospital, Frankfurt, Germany
Locations (33):
- Austria (4):
  - Bezirkskrankenhaus Hall, Hall in Tirol
  - Medizinische Universität Innsbruck, Innsbruck
  - Bezirkskrankenhaus Kufstein, Kufstein
  - St. Vinzenz Krankenhaus Zams, Zams
- Germany (29):
  - Klinikum Altenburger Land GmbH, Altenburg
  - Gesundheitszentrum St. Marien GmbH am Klinikum St. Marien, Amberg
  - Studienzentrum f. Hämatologie, Onkologie u. Diabetologie, Aschaffenburg
  - Klinikum Bayreuth, Bayreuth
  - Praxis Onkologie, Cologne
  - Klinikum Dortmund GmbH, Dortmund
  - Universitätsklinik Dresden, Dresden
  - Westdeutsches Tumorzentrum - Universitätsklinikum Essen, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - MVZ Onkologische Schwerpunktpraxis, Frankfurt
  - Klinikum der Johann Wolfgang-Universität Frankfurt, Frankfurt a.M.
  - Martin-Luther Universität Halle, Halle
  - Onkologische Schwerpunktpraxis, Hamburg
  - Universitätsklinkum Heidelberg - Nationales Centrum f. Tumorerkrankungen, Heidelberg
  - Marienhospital Herne, Herne
  - Onkologische Schwerpunktpraxis, Hildesheim
  - Onkologische Schwerpunktpraxis, Hof
  - Praxis für Hämatologie und internistische Onkologie, Kronach
  - Klinikum der Stadt Ludwigshafen, Ludwigshafen
  - Klinikum Lüdenscheid, Lüdenscheid
  - Klinikum Magdeburg gGmbH, Magdeburg
  - Johanness-Gutenberg Universität Mainz, Mainz
  - Praxis für Hämatologie und internistische Onkologie, München
  - Gemeinschaftspraxis f. Hämatologie u. Onkologie, Münster
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Prosper-Hospital, Recklinghausen
  - Onkologische Schwerpunktpraxis, Hämatologie und Onkologie, Trier
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Nordoberpfalz AG, Weiden Oberpfalz